CLINICAL TRIAL: NCT02029183
Title: Screening and Treatment of in Sleep Apnea Hypopnea Syndrome（SAHS)Patients With Acute Ischemic Stroke
Brief Title: Screening and Treatment of SAHS in Patients With Acute Ischemic Stroke
Acronym: SAHS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Dongsheng Fan, Professor, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2694-01
Record Dates: First submitted 2013-11-17; First posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Ischemic Stroke; Sleep Apnea Syndrome
Keywords: stroke, SAHS, BiPAP
MeSH Terms: conditions — Ischemic Stroke; Sleep Apnea Syndromes; Stroke; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bi-level positive airway pressure (Experimental): bi-level positive airway pressure for 6 hour per night，total 7 days
  Interventions: Device: Bi level positive pressure ventilation; Device: bi-level positive airway pressure

INTERVENTIONS:
Device: Bi level positive pressure ventilation — Bi level positive pressure ventilation should be given for subject for 6 hours per night ，total 7 times.
Device: bi-level positive airway pressure

SUMMARY:
Ischemic stroke is a kind of common disease with great harm. In acute stage of stroke there is sharply increasing morbidity of sleep apnea hypopnea syndrome. Our suppose that treatment with noninvasive ventilation for patients with acute ischemic stroke should improve the functional prognosis（measuring with 90d modified Rankin score）.

DETAILED DESCRIPTION:
In acute state of ischemic stroke，if patients with sleep apnea hypopnea syndrome may need additional respiratory management such bi-level positive airway pressure.We supposed the patients with stroke can take benefit of functional recovery form bi-level positive airway pressure. We choose the patients who suffered ischemic stroke in 48 hours ，then evaluate the respiratory status. Stroke patients who were diagnosed as sleep apnea hypopnea syndrome will accept additional treatment with bi-level positive airway pressure for 7 night（per night 6 hours）.Then the modified Rankin scale score and NIHSS will be recorded at 30 days and 90 days after stroke.

ELIGIBILITY:
Inclusion Criteria:

* ischeic stroke onset within 48 hours , NIHSS:4-15

Exclusion Criteria:

* mRs>2 before onset of enrollment severe hepatic renal insufficiency cancer in reached an advanced stage

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale score | 90 days after symptoms
  0-2 Modified Rankin Scale score should be recognized good functional prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, P, Study Chair — Peking University Third Hospital
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China